CLINICAL TRIAL: NCT06833801
Title: Application of Intelligent Care Systems in Radiation Therapy: Enhancing Patient Safety and Reducing Anxiety Through System Optimization, Enhanced Education Strategies, and Real-Time Blood Data Monitoring
Brief Title: Application of Intelligent Care Systems in Radiation Therapy: Enhancing Patient Safety and Reducing Anxiety Through System Optimization and Real-Time Blood Data Monitoring
Acronym: ICS-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-A-031
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Radiation Therapy; Chemoradiotherapy; Anxiety; Adherence
Keywords: Radiation Therapy; Intelligent Care System; Real-Time Blood Data Monitoring; Patient Safety; Oncology Treatment Compliance; Cancer Treatment Anxiety; Clinical Decision Support System; Health Education in Radiation Oncology; Automated Blood Test Alerts; Supportive Care in Cancer Patients
MeSH Terms: conditions — Anxiety Disorders | interventions — Caffeine; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This study involves two parallel groups:
  Intervention Group - Receives real-time blood monitoring alerts, enhanced patient education materials, and internal warning reminders.
  Control Group - Receives standard care without system enhancements.
Who Masked: Participant
Masking Description: Participants will not be informed of the specific intervention details, but healthcare providers and researchers will be aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intelligent Care System Group (Intervention Group) (Experimental): Participants in this group will receive an optimized intelligent care system designed to enhance patient safety, improve treatment adherence, and reduce anxiety during radiation therapy. This system includes real-time blood data monitoring alerts, enhanced patient education materials, and internal warning reminders.
  Interventions: Device: Real-Time Blood Data Monitoring System (Device/Software Integration); Behavioral: Enhanced Patient Education Materials (Behavioral/Educational Intervention); Behavioral: Internal Warning Signs and Alerts (Behavioral Intervention)
- Standard Care Group (Control Group) (No Intervention): Participants in this group will receive standard care without the optimized intelligent care system interventions. They will continue their treatment following existing clinical practices without additional automated monitoring or enhanced education strategies.

INTERVENTIONS:
Device: Real-Time Blood Data Monitoring System (Device/Software Integration) — Description: An alert function will be integrated into the hospital's electronic system, allowing healthcare providers to view real-time blood test results of radiation therapy patients. The system will notify both medical staff and patients of abnormal results, prompting timely intervention.
  Mode of Delivery: Hospital Information System (HIS) Integration Purpose: Improve treatment safety by reducing delays in managing abnormal blood counts.
  Arms: Intelligent Care System Group (Intervention Group)
Behavioral: Enhanced Patient Education Materials (Behavioral/Educational Intervention) — Description: Optimized educational pamphlets and multimedia resources will be provided to patients, including clear self-care instructions and guidance on reporting blood test needs during radiation therapy.
  Mode of Delivery: Printed materials, multimedia resources, verbal education by medical staff Purpose: Improve patient understanding and engagement in their treatment process.
  Arms: Intelligent Care System Group (Intervention Group)
Behavioral: Internal Warning Signs and Alerts (Behavioral Intervention) — Description: Physical reminder signs will be placed in high-traffic patient areas (e.g., check-in counters, treatment rooms) to prompt patients to report discomfort or abnormal symptoms, especially related to blood test needs.
  Mode of Delivery: Visual reminders placed within the radiation oncology department Purpose: Increase patient awareness and adherence to treatment safety protocols.
  Arms: Intelligent Care System Group (Intervention Group)

SUMMARY:
This study aims to evaluate the impact of an intelligent care system on radiation therapy patients, focusing on real-time blood data monitoring, optimized patient education, and internal alert systems. The goal is to enhance patient safety, improve treatment adherence, and reduce anxiety by integrating an alert function into the hospital's existing system.

Key interventions include:

Real-time blood monitoring alerts: Healthcare providers will receive automatic notifications of abnormal blood test results to ensure timely intervention.

Optimized patient education materials: Clearer guidance will help patients proactively communicate blood test needs and manage their health during radiation therapy.

Internal reminders: Visual signs and alerts in treatment areas will reinforce patient awareness and engagement.

The study will compare patients receiving these interventions with those under standard care, assessing treatment compliance, anxiety levels, and clinical outcomes over a 12-month period.

DETAILED DESCRIPTION:
Background & Rationale Cancer patients undergoing radiation therapy often experience changes in blood cell counts, particularly when combined with chemotherapy, affecting treatment safety and completion rates. Lack of real-time monitoring and patient engagement can lead to delays or complications in treatment. This study integrates an intelligent care system into clinical practice to enhance patient monitoring and education, reducing treatment interruptions and improving outcomes.

Study Objectives

System Optimization: Develop an automated blood data monitoring system that alerts medical staff and patients about abnormal results.

Patient Education Enhancement: Improve educational materials to guide patients on self-care and timely communication with healthcare providers.

Internal Warning Implementation: Install reminder signs in treatment areas to increase awareness and compliance.

Study Design

Type: Interventional (Clinical Trial) Design: Randomized, parallel assignment

Groups:

Intervention Group: Receives real-time monitoring alerts, enhanced education materials, and internal warning systems.

Control Group: Receives standard care without system enhancements. Primary Outcomes: Anxiety reduction (measured by BSRS-5) and treatment adherence rates.

Secondary Outcomes: Blood data changes, patient understanding of self-care, and clinical treatment outcomes.

Expected Impact By combining real-time data monitoring with patient education and engagement, this study aims to create a safer, more informed treatment experience, reducing patient anxiety and enhancing overall treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiation therapy combined with chemotherapy.
* Age ≥ 18 years.
* Ability to understand and comply with the study protocol.
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Patients with severe cognitive impairment or intellectual disability, affecting their ability to understand or follow study procedures.
* Patients unwilling to complete study questionnaires.
* Any mental health condition (e.g., major depressive disorder, severe anxiety disorder) that could interfere with participation.
* Patients with conditions requiring immediate intervention that would make study participation impractical.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Anxiety Levels During Radiation Therapy | Baseline (before radiation therapy) and 3 weeks after treatment initiation
  The study will measure changes in patient anxiety levels before and after the intervention using the Brief Symptom Rating Scale-5 (BSRS-5). The BSRS-5 is a validated psychological assessment tool designed to screen for psychological distress, including anxiety, depression, hostility, interpersonal sensitivity, and insomnia.
  Scale Range: The BSRS-5 consists of five items, each scored from 0 (not at all) to 4 (extremely severe).
  Minimum Score: 0 (indicating no psychological distress). Maximum Score: 20 (indicating severe psychological distress). Interpretation: Higher scores indicate worse psychological distress. Outcome Goal: A decrease in BSRS-5 scores in the intervention group compared to the control group will indicate reduced anxiety and improved psychological well-being.
Treatment Adherence Rate During Radiation Therapy | Throughout the entire course of radiation therapy (typically 4-6 weeks)
  The study will track patient compliance with the prescribed radiation therapy regimen. Compliance will be measured through attendance records, completion of scheduled treatment sessions, and physician assessments. The intelligent care system is expected to improve adherence by increasing patient engagement and awareness through automated alerts and improved educational materials. A higher completion rate in the intervention group compared to the control group will indicate improved treatment adherence.

SECONDARY OUTCOMES:
Change in Blood Cell Counts During Radiation Therapy | Weekly from baseline (Week 0) until treatment completion (approximately 4 to 6 weeks).
  This study will evaluate how often abnormal blood cell counts (White Blood Cell [WBC], Hemoglobin [Hb], and Platelet [PLT] levels) are detected and addressed using the real-time blood data monitoring system. The system provides timely alerts for abnormal values, enabling healthcare providers to intervene promptly.
  Assessment Tool: Electronic medical records of routine blood test results. Outcome Goal: The intervention group is expected to have fewer missed abnormal results and faster clinical response times compared to the control group, indicating improved patient safety.
Patient Understanding of Self-Care and Blood Test Needs | Pre-treatment and after 3 weeks of treatment
  Assess patient awareness and knowledge of self-care practices and the importance of blood test monitoring during radiation therapy. Patients will receive optimized educational materials, and their understanding will be evaluated through a self-reported questionnaire. A higher score in the intervention group compared to the control group will indicate improved patient education and awareness.
Patient Satisfaction with the Intelligent Care System | At Week 6 (end of radiation therapy treatment, typically 4 to 6 weeks after initiation).
  Measure patient satisfaction regarding the new real-time blood monitoring alerts and enhanced educational materials provided as part of the intelligent care system. A patient-reported satisfaction survey will be conducted to evaluate the perceived usefulness and acceptability of the system.
  Assessment Tool: Patient-reported satisfaction survey. Outcome Goal: Higher satisfaction scores in the intervention group compared to the control group, indicating greater patient acceptance and perceived benefits of the system.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No